CLINICAL TRIAL: NCT06523842
Title: Cross Culture Adaptation Validity and Reliability of Arabic Version of Cornell Muscloskeletal Discomfort Questionnaire
Status: Enrolling by invitation | Type: Observational
Sponsor: Sara Mortada Mohamed (Other)
Responsible Party: Sponsor-Investigator, Sara Mortada Mohamed, demonstrator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 012/0040111
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Translation of Cornell Muscloskeletal Questionnair Into Arabic Language
Keywords: arabic version of cornell muscloskeletal questionnaire; validity and reliability
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire — cronell questionnaire for assessment muscloskeletal discomfort in sedentary and standing workers males and females

SUMMARY:
The purpose of this study is to translate and test face validity,content validity, Feasibility, internal consistency reliability and Test retest reliability of adapted Arabic-language version of Cornell musculoskeletal discomfort questionnaires in patients with musculoskeletal

DETAILED DESCRIPTION:
1.Study design: This study is a prospective observational study; it follows the recommendations of to test (face, content and construct) validity, feasibility, and (internal consistency and test re-test) reliability

.Participants: To have a good sample size researchers preferred to have a multiplier of 10, so as the RC-QOL questionnaire contains 54 questions, so the number of participants was 54 x10 =540 Methods The Cornell Musculoskeletal Discomfort Questionnaire is a 54-item questionnaire containing a body map diagram and questions about the prevalence of musculoskeletal ache, pain or discomfort in 18 regions of the body during the previous week .The Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) are a set of tools developed by Dr. Alan Hedge and his team at Cornell University. They are designed to assess musculoskeletal discomfort among office workers and other populations. .The CMDQ includes different versions for sedentary and standing workers, as well as specific questionnaires for hand discomfort Scoring Guidelines - Cornell Musculoskeletal and Hand Discomfort Questionnaires

These questionnaires are for research screening purposes and not for diagnostic purposes. Scores can be analyzed in 4 ways:

1. by simply counting the number of symptoms per person
2. by summing the rating values for each person
3. by weighting the rating scores to more easily identify the most serious problems as follows: Never = 0 1-2 times/week = 1.5 3-4 times/week = 3.5 Every day = 5 Several times every day = 10
4. by multiplying the above Frequency score (0,1.5 , 3.5, 5, 10) by the Discomfort score (1,2,3) by the Interference score (1,2,3) In the computational analyses missing values can be coded as 0. If the missing value is for the frequency score then use this as a zero in multiplying, i.e. all combinations of Frequency, Discomfort and Interference become 0. However, if the missing value is in the Discomfort or Frequency score then treat it as missing so that the multiplied score will be at least the value of the Frequency score.

The individual items should also be analyzed to determine where there may be a postural problem for the person.

Translation Process and the Adaptation of Instruments (Assessment Tool) into The Arabic Language:

Translation is merely the first stage of the adaptation process. When adapting an instrument, cultural, idiomatic, linguistic and contextual aspects concerning its translation should be considered Once the instrument is adapted, studies between different populations that compare the characteristics of individuals in different cultural contexts may be conducted. Accordingly, research on the adaptation of instruments has placed great emphasis on comparing results through studies that use different samples .

The instrument adaptation entails six essential stages:

1. Instruments translation from the source language into the target language,
2. Synthesis of the translated versions,
3. Analysis of the synthesized version by expert judges,
4. Instrument evaluation by the
5. Target population,
6. Back translation, and
7. A pilot study

Stages of the Translation Process and the Adaptation of Instruments Instrument Translation into the New Language:

When adapting an instrument, one must first consider its translation from the source language into the target language, that is, the language with which the new version will be used. This is a complex process and requires tremendous care to ensure that the final version is not only suitable for the new context but is also consistent with the original version. Therefore, an appropriate translation requires a balanced treatment of linguistic, cultural, contextual, and scientific information .

Ergonomic assessment is commonly used to identify hazards in the work environment and to suggest ways to lessen them . Useful ergonomic assessment tools include: Rapid Entire Body Assessment (REBA) through observation and the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) through a questionnaire.

The research consensus in this area suggests that independent, bilingual translators should be summoned to adapt the items into the new language . Although a single translator was previously believed to be suitable for the completion of the translation process, the presence of at least two bilingual translators is now recommended for completing this process, thereby minimizing the risk of linguistic, psychological, cultural,and both theoretical and practical understanding biases .

Many suggestions for translation focus on the quality of the translators. For example, Hambleton (2005) argues that translators should be fully proficient in both languages of interest and familiar with the cultures associated with the respective languages of each group.

Beaton et al. (2000) advocate that translators must be fluent in the source language of the instrument and native in the target language. Such characteristics enable the translation process to consider the nuances of the language for which the instrument is intended, which ensures a greater cultural fit of the adaptation process .

One of the translators should be familiar with the assessed construct, while a second translator should not be aware of the translation goals. The first translator's adaptation tends to provide a higher scientific similarity of the instrument, which delivers a higher equivalence from a psychometric perspective. Conversely, the second translator's adaptation tends to show a lower probability of deviation concerning the meaning of items. The second translator tends to offer a version that best reflects the language used by the target population because he or she is less influenced by the academic purpose of the translation .

Synthesis of the Translated Versions:

After the process of instrument translation from the source language into the target language, the researcher should have at least two versions of the translated instrument. At this stage, the process of summarizing both versions begins. Summarizing the versions of an instrument means that the researcher compares the different translations and assesses their semantic, idiomatic, conceptual, linguistic and contextual differences, with the sole purpose of creating a single version.

During this process, it is common to identify two possible sources of complications:

1. Complex translations that may hinder the understanding of the population for whom the instrument is intended.
2. Overly simplistic translations that underestimate the item content. The evaluation of different translations of an instrument should be conducted for each item separately. Throughout this process, the committee (judges and authors) should assess the compatibility between the translated versions and the original instrument

The choice of which version to use must be made through consensus among the judges, and never by imposition . When possible, an external observer should be prompted to transcribe the entire synthesis process, especially regarding the choice of items to be used . This transcription provides a qualitative overview of the process to the researcher. At the end of this stage, the researcher will hold a single version of the instrument, which may include items translated by one or more than one translators .

Evaluation of the Synthesized Version by Experts:

After the synthesis of translated versions has been finished, the researcher should still rely on the help of a committee of either experts in the area of psychological evaluation or on those with specific knowledge of what the instrument assesses. These experts will assess other important aspects, such as the structure, layout, instrument instructions, and both the scope and adequacy of expressions contained in the items .

The experts will then consider, for example, whether the terms or expressions may be generalized for different contexts and populations (that is, different regions of a given country) and whether the expressions are a good fit for the population for whom the instrument is intended. Aspects of the instrument layout will also be analyzed because they are as indispensable as the linguistic aspects of the items, especially regarding the instruments to be used on specific populations, including children and the elderly. The clarity of the content, the suitability of font formats and sizes, the arrangement of information on the instrument, are also analyzed .

Translation, synthesis and evaluation of the translated version are the first steps in the instrument's adaptation into a new culture. After completing these stages, the first version of the instrument will be ready for the next stage: instrument evaluation by the target population.

Evaluation by the Target Population:

This stage of the process aims to verify whether the items, the response scale and the instructions are comprehensible for the target population. Thus, this procedure aims to investigate whether the instructions are clear, whether the terms found in the items are appropriate, whether the expressions correspond to those used by the group, and other aspects. The subjects who participate in this step may vary depending on the characteristics of the respondents for whom the instrument is intended .

Back-Translation:

Back-translation is also suggested as an additional quality control check . From our perspective, this procedure must follow all semantic and idiomatic adjustment procedures because the instrument must be -ready‖ for final evaluation by the original author. Back-translation refers to translating the synthesized and revised versions of the instrument into the source language. Its aim is to evaluate the extent to which the translated version reflects the item content of the original version. Back-translation must be performed by at least two translators other than those who performed the first translation .

The purpose of back-translation, however, should not be a literal interpretation of the original version and the translated versions. Instead, the back-translation process should be used as a tool to identify words that were not clear in the target language and to identify inconsistencies or conceptual errors in the final version. Back-translation may also be used as a practical tool so that the researcher who is adapting the instrument may communicate with the author of the original instrument. When the author has access to the back-translated version of the instrument, the author may state whether the items share the same meanings as those of the original items .

Pilot Study:

Before claiming that a new instrument is ready for application, one must perform a pilot study. The pilot study refers to a previous application of the instrument in a small sample that reflects the sample/target-population characteristics. Once again, the appropriateness of items regarding their meaning and difficulty, in addition to instructions for conducting the test, should be assessed during this process .

After considering the modifications suggested in the first pilot study, a second pilot study (or as many as needed) is necessary to assess whether the instrument is ready to be used. To avoid any type of bias, the changes suggested by the pilot study (or studies) should be implemented with the help of a committee of experts and should never be performed solely by the field researcher .

ELIGIBILITY:
Inclusion Criteria:

- Male and female

* Being sedentary office workers
* Being standing workers .Being literate and speaking Arabic. .Patients were aged from 18 to 60 years old.

Exclusion Criteria:

* Inability to complete the form due to cognitive impairment. .Individuals who were unable or unwilling to complete study outcomes or provide informed consent.
* Systematic inflammatory rheumatic diseases .Neurological conditions. .Psychiatric disorders.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: male and female sedentary and standing workers
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-29 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
cronell muscloskeletal discomfort questionnaire | 15 minutes
  questionnaire for assessment muscloskeletal discomfort in sedentary and standing workers in previous weeks How can I classify the severity of discomfort into mild, moderate, or more. The discomfort score is a severity of discomfort. Originally we had it as 'mild', 'moderate' and 'severe discomfort', but we found that people more easily understood the categories 'slightly', 'moderately' and 'very uncomfortable' . if you like you can replace the scale point titles with 'mild', 'moderate' and 'severe discomfort

CONTACTS AND LOCATIONS:
Overall Officials: haitham El Hafez, prof, Study Director — cairo university ,egypt
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided